CLINICAL TRIAL: NCT07360704
Title: Genotypes and Craniofacial Phenotypes in Orthodontic Patients With Marfan and Loeys-Dietz Syndromes: Observational Retrospective Study
Brief Title: Genotypes and Craniofacial Phenotypes in Orthodontic Patients With Marfan and Loeys-Dietz Syndromes
Status: Completed | Type: Observational
Sponsor: Andrea Scribante (Other)
Responsible Party: Sponsor-Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Organization: University of Pavia (Other)
Other Study IDs: 2026-MARFANLDS
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Marfan Syndrome; Loeys-Dietz Syndrome
MeSH Terms: conditions — Marfan Syndrome; Loeys-Dietz Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- FBN1Cys (Marfan syndrome, cysteine missense variants): This arm included patients diagnosed with Marfan syndrome carrying missense variants affecting cysteine residues of the FBN1 gene.
  Interventions: Diagnostic Test: Cephalometric analysis
- FBN1m (Marfan syndrome, non-cysteine missense variants): This arm comprised patients with Marfan syndrome carrying missense FBN1 variants not involving cysteine residues.
  Interventions: Diagnostic Test: Cephalometric analysis
- FBN1tp (Marfan syndrome, truncating variants): Patients in this arm were affected by Marfan syndrome and carried truncating FBN1 variants, including nonsense, frameshift, or splicing mutations.
  Interventions: Diagnostic Test: Cephalometric analysis
- LD (Loeys-Dietz syndrome): This arm included patients diagnosed with Loeys-Dietz syndrome carrying pathogenic variants in TGFBR1 or TGFBR2 genes.
  Interventions: Diagnostic Test: Cephalometric analysis
- Control group: A control group matched for age and sex was added for all syndromic patients.
  Interventions: Diagnostic Test: Cephalometric analysis

INTERVENTIONS:
Diagnostic Test: Cephalometric analysis — Lateral cephalometric radiographs with cephalometric tracings were performed to evaluate craniofacial patterns.

SUMMARY:
The aim of this retrospective observational study is to investigate the association between genotype and craniofacial phenotype in orthodontic patients affected by Marfan and Loeys-Dietz syndromes. A total of 39 patients aged between 4 and 18 years were enrolled and stratified into four groups according to the underlying pathogenic genetic variants. Lateral cephalometric radiographs were analyzed to assess sagittal, vertical, and cranial base skeletal relationships. Each patient group was compared with age- and sex-matched controls, as well as between syndromes and among Marfan subgroups. Statistical analyses were performed to evaluate differences in craniofacial parameters and to explore potential genotype-phenotype correlations relevant for orthodontic diagnosis.

DETAILED DESCRIPTION:
This retrospective observational study aims to investigate the association between genotype and craniofacial phenotypic variation in orthodontic patients affected by Marfan syndrome (MFS) and Loeys-Dietz syndrome (LDS). Patients aged between 4 and 18 years who referred to the Unit of Orthodontics and Paediatric Dentistry and had a confirmed genetic diagnosis were considered eligible for inclusion. Parents or legal guardians provided informed consent prior to data collection.

A total of 39 patients were enrolled and divided into four groups according to the underlying pathogenic genetic variant:

* Group FBN1Cys: Marfan patients with missense cysteine variants of the FBN1 gene.
* Group FBN1m: Marfan patients with missense non-cysteine variants of the FBN1 gene.
* Group FBN1tp: Marfan patients with truncating FBN1 variants (nonsense, frameshift or splicing mutations).
* Group LD: Patients with Loeys-Dietz syndrome carrying pathogenic variants in TGFBR1 or TGFBR2 genes.

An age- and sex-matched control group without genetic disorders and without previous orthodontic treatment was selected for each study group. All patients underwent orthodontic diagnostic records including lateral cephalometric radiographs. Due to the retrospective nature of the study and the use of different radiographic units, only angular cephalometric measurements were considered.

Cephalometric analysis was performed using dedicated software according to Giannì's method, evaluating sagittal, vertical and cranial base relationships. Each patient was compared with the corresponding control group, between MFS and LDS patients, and among the Marfan subgroups. All measurements were performed by a single operator and intra-rater reliability was assessed.

Sample size was defined by the availability of patients affected by these rare genetic disorders who met the inclusion criteria during the study period. Descriptive statistics were calculated for all cephalometric parameters. Shapiro-Wilk test was applied to assess data normality. Differences between groups were evaluated using ANOVA, followed by Tukey's post-hoc test when appropriate.

Statistical analysis was conducted using R software, with significance for all tests predetermined at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Marfan/Loeys-Dietz syndrome;
* formal request of parents or legal guardians for orthodontic evaluation;
* aged between 4 and 18;
* no previous orthopaedic or orthodontic treatment.

Exclusion Criteria:

* History of craniofacial anomalies (e.g., cleft lip/palate, craniosynostosis) or syndromic conditions other than Marfan/Loeys-Dietz syndrome;
* previous orthopaedic or orthodontic treatment;
* poor quality cephalograms.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients referring for orthodontic consultation from the Unit Centre for Inherited Cardiovascular Diseases, IRCCS Foundation, University Hospital Policlinico San Matteo, Pavia, Italy
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-07-07 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
ANB angle | Baseline
  The ANB angle will be measured on lateral cephalometric radiographs to assess the sagittal skeletal relationship between the maxilla and mandible. Comparisons will be performed between genotype-based case groups and age- and sex-matched controls, as well as among case groups when applicable.

SECONDARY OUTCOMES:
SNA angle | Baseline
  SNA angle will be measured to assess maxillary position relative to the cranial base.
SNB angle | Baseline
  SNB angle will be measured to assess mandibular position relative to the cranial base.
Vertical skeletal pattern (SN-MP angle) | Baseline
  SN-MP angle will be measured to evaluate mandibular plane inclination and vertical skeletal pattern.
Intermaxillary vertical relationship (PP-MP angle) | Baseline
  PP-MP angle will be measured to assess vertical discrepancy between the palatal plane and the mandibular plane.
Occlusal plane relationships (Occ-MP and Occ-PP angles) | Baseline
  Occ-MP and Occ-PP angles will be measured to assess occlusal plane inclination relative to the mandibular and palatal planes.
Cranial base morphology (N-S-Ar and S-Ar-Go angles) | Baseline
  N-S-Ar and S-Ar-Go angles will be measured to evaluate cranial base flexure and posterior cranial base-mandibular ramus relationship.
Mandibular morphology (Ar-Go-N angle) | Baseline
  Ar-Go-N angle will be measured to assess mandibular morphology and angular configuration.
Facial vertical pattern (N-Go-Gn angle) | Baseline
  N-Go-Gn angle will be measured to assess facial vertical growth pattern.
Maxillary incisor inclination (11-Occ and 11-PP) | Baseline
  11-Occ and 11-PP measurements will be used to assess maxillary central incisor inclination relative to the occlusal and palatal planes.
Mandibular incisor inclination (41-Occ and 41-MP) | Baseline
  41-Occ and 41-MP measurements will be used to assess mandibular central incisor inclination relative to the occlusal and mandibular planes.
Nasolabial angle (NLA) | Baseline
  The nasolabial angle will be measured to assess soft tissue profile characteristics.
Facial angle (FA) | Baseline
  The facial angle will be measured to evaluate overall facial profile morphology.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — Associate Professor, Principal Investigator
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.